CLINICAL TRIAL: NCT07093645
Title: Promoting Well-being Among European Adolescents - an Inclusive and Digital Program to Strengthen Social-emotional Competences (SEL4@ll)
Brief Title: Serious Game-Based School Intervention to Enhance Socio-Emotional Competence and Well-Being in European Adolescents
Acronym: SEL4@ll
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: Universitat Politècnica de València (Other); University Of Perugia (Other); University of Eastern Finland (Other); University of Greifswald (Other); European Union (Other)
Responsible Party: Principal Investigator, Konstanze Schoeps, Associate Professor of Personality, Evaluation and Psychological Treatments, University of Valencia
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024-PSILOG-3715935; KA220-MV-22-36-89514 (Other Grant/Funding Number: European Union)
Record Dates: First submitted 2025-05-16; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: None - Study is to Determine Safety in Healthy Participants
Keywords: socioemotional competences; inclusion; adolescence; well-being; school well-being; student burnout
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: There are two groups: one experimental and one control. The experimental group will play the game and undergo pre- and post-game evaluations, as well as an impact evaluation some time after playing. The control group will undergo the same evaluations and will be offered the game as a reward.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Playing serious game and using didactic material at school (Experimental): The experimental group will play the game and complete pre- and post-game evaluations, as well as a follow-up impact assessment. This will help assess the game's effectiveness in improving socio-emotional competencies and overall well-being.
  Interventions: Device: SEL4@ll
- Only assessment with serious games as the reward (No Intervention): The control group will undergo the same evaluations as the experimental group, but will not play the game. They will receive the game as a reward after completing the assessments, allowing for a comparison of results between the two groups.

INTERVENTIONS:
Device: SEL4@ll — SEL4@ll is a school-based digital intervention targeting students aged 10-16 (Primary and Secondary Education). It combines: (1) a serious game with five missions promoting SEL skills (1/week), playable online at home or school; (2) a digital teacher handbook with classroom activities used 1-2 times per week; and (3) online surveys to assess impact. The program lasts 8 weeks: 2 weeks for pre/post assessments and 6 weeks of gameplay and classroom sessions. Surveys are administered online (3 waves), and optional focus groups are conducted with a subsample of students. Teachers complete an online evaluation after implementation.
  Arms: Playing serious game and using didactic material at school

SUMMARY:
The goal of this study is to evaluate whether a digital, game-based social-emotional education intervention (SEL4@ll) can improve socio-emotional competencies, well-being, and inclusion in primary and secondary school students aged 10-16 across four European countries. The main questions it aims to answer are:

* Does participating in the SEL4@ll serious game increase students' socio-emotional competencies, such as self-awareness, empathy, and decision-making?
* Does the program enhance students' sense of well-being and social inclusion within the classroom environment?

Researchers will compare outcomes between students who participate in the SEL4@ll intervention and those in the control group who follow standard curricular activities to see if the game-based program leads to significant improvements.

Participants will:

* Play a serious game focused on five themed "portals" that develop emotional intelligence, leadership, gratitude, resilience, and justice.
* Complete questionnaires at three different time points (pre-, post-, and follow-up) to assess changes in competencies.
* Take part in focus groups (students) and provide implementation feedback (teachers).
* Engage in teacher-led activities and worksheets designed to support reflection and integration of SEL4@ll content.

DETAILED DESCRIPTION:
SEL4@ll is an EU-funded, cross-national intervention designed to promote social-emotional learning (SEL) among primary and secondary school children using a serious game supported by pedagogical resources. The intervention aligns with the Collaborative for Academic, Social, and Emotional Learning (CASEL) framework and draws on evidence-based models of SEL, life skills development, character education, and positive youth development.

The serious game is the centerpiece of the intervention and is structured around five narrative "gates or portals," each of which targets three interrelated competencies:

Gate of Self: sense of meaning, resilience, leadership

Gate of Emotion: emotional intelligence, empathy, compassion

Gate of People: communication, gratitude, positive influence

Gate of Knowledge: motivation, growth mindset, critical thinking

Final Mission: equality, responsibility, justice

The game presents students as protagonists navigating magical environments to overcome a symbolic "dark force" by mastering SEL competencies, represented as branches of a "skill tree." The game is hosted online, accessible through a browser, and available in English, Spanish, Italian, German, and Finnish.

To facilitate educational integration, SEL4@ll provides a digital teacher handbook and didactic materials-including lesson plans and reflection worksheets-that help structure learning around the game content. Teachers play a vital role by guiding discussions and activities before and after gameplay.

The evaluation strategy includes both quantitative and qualitative components and follows a co-creation approach:

A three-wave design assesses students' development over time (pre-test, post-test, and delayed follow-up).

Quantitative measures include validated self-report questionnaires focused on SEL competencies, well-being, and perceived social inclusion.

Qualitative data are gathered through student focus groups and teacher interviews to explore experiences, perceptions, and implementation barriers.

Feedback from critical friends and stakeholders is used to iteratively refine the program materials and processes.

This study is conducted simultaneously in Germany, Spain, Italy, and Finland, allowing for a robust cross-cultural analysis of the intervention's effectiveness. Data will be analyzed both within and across countries to identify universal impacts and culturally specific outcomes, thereby informing future adaptation and scalability of the SEL4@ll model in broader European educational contexts.

This study is part of the Erasmus+ project "Promoting well-being among European adolescents: An inclusive and digital programme to strengthen socio-emotional competencies - SEL4@ll" and aims to contribute to evidence-based innovation in the transition form primary to secondary education by leveraging digital tools and inclusive pedagogy.

ELIGIBILITY:
Inclusion Criteria

Participants must meet all of the following criteria to be included in the study:

* Be within the target age range (typically 10-16 years old, corresponding to 5th-6th grade of primary or 1st-4th year of secondary education).
* Have written informed consent provided by a parent or legal guardian.
* Complete all three measurement points (pre-test, post-test, and follow-up assessments).
* Attend school regularly (i.e., not chronically absent).

Exclusion Criteria

Participants will be excluded from the study if they:

* Do not obtain parental/legal guardian consent.
* Have significant cognitive, developmental, or language impairments that prevent them from understanding or completing the intervention or assessment tools.
* Are absent for a prolonged period during the implementation phase (e.g., due to illness, transfer, or other reasons).
* Participate in another intervention targeting similar outcomes during the study period, which may confound results.

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Social Skills Improvement System Social and Emotional Learning Brief Scales (Anthony et al., 2020) | Three measurement points: T1 (one week before intervention "baseline"), T2 (after intervention, eight weeks after T1) and T3 (follow-up, three months after T1).
  The SSIS SEL Brief Scales is a 20-item questionnaire developed to assess social and emotional learning (SEL) competencies in children and adolescents. The items are organized into five domains that align with the core SEL areas defined by the CASEL framework (2020): self-awareness, self-management, social awareness, relationship skills, and responsible decision-making. Each item is rated on a 4-point Likert scale, from 1 (Not True) to 4 (Very True), resulting in a total score ranging from 20 (minimum) to 80 (maximum). Higher scores reflect stronger perceived social and emotional competencies.

SECONDARY OUTCOMES:
Questionnaire about student well-being (Hascher et al., 2018) | Three measurement points: T1 (one week before intervention "baseline"), T2 (after intervention, eight weeks after T1) and T3 (follow-up, three months after T1).
  The questionnaire consists of 19 items rated on a 6-point Likert scale ranging from 1 (Never) to 6 (Very Often), and is designed to assess six dimensions of student well-being: positive attitudes toward school, enjoyment in school, worries in school, physical complaints in school, social problems in school, and positive academic self-concept. Each dimension is measured with three items, resulting in a minimum score of 3 and a maximum score of 18 per scale.
  Three of the dimensions-positive attitudes toward school, enjoyment in school, and positive academic self-concept-are positive indicators, where higher scores reflect higher levels of well-being. The other three dimensions-worries in school, physical complaints in school, and social problems in school-are negative indicators, where higher scores indicate lower levels of well-being.
Perception of Inclusion Questionnaire (Venetz et al., 2015) | Three measurement points: T1 (one week before intervention "baseline"), T2 (after intervention, eight weeks after T1) and T3 (follow-up, three months after T1).
  The questionnaire consists of 12 items rated on a 4-point Likert scale, ranging from 1 (Not at all true) to 4 (Certainly true). It measures three key aspects of students' social inclusion at school: emotional self-inclusion (feeling accepted and valued), social inclusion (feeling part of the peer group), and academic self-concept (perception of one's own academic competence). Each dimension is assessed through four items, resulting in a minimum score of 4 and a maximum score of 16 per subscale, and a total score ranging from 12 (minimum) to 48 (maximum).
  Higher scores reflect greater levels of perceived inclusion, indicating that the student feels more emotionally connected, socially integrated, and academically competent within the school environment.

CONTACTS AND LOCATIONS:
Overall Officials: Konstanze Schoeps, Principal Investigator — University of Valencia
Locations (1):
- University of Valencia, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schoeps K, Postigo-Zegarra S, Signorelli A, Morganti A, Lozano-Quilis JA, Hoferichter F. SEL4@ll program for social and emotional development among European adolescents: a study protocol for a randomized controlled trial. BMC Psychol. 2025 Nov 28;13(1):1318. doi: 10.1186/s40359-025-03678-w. PMID 41316371